CLINICAL TRIAL: NCT00395135
Title: BLOOM: Behavioral Modification and Lorcaserin for Overweight and Obesity Management; A 104-Week, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Safety and Efficacy of Lorcaserin Hydrochloride in Obese Patients
Brief Title: BLOOM: Behavioral Modification and Lorcaserin for Overweight and Obesity Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APD356-009
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2013-01

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; lorcaserin; APD356; BLOOM; Hypertension; Dyslipidemia; Sleep apnea; glucose tolerance; cardiovascular disease; Arena
MeSH Terms: conditions — Obesity; Weight Loss; Hypertension; Dyslipidemias; Sleep Apnea Syndromes; Cardiovascular Diseases | interventions — lorcaserin; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lorcaserin 10 mg BID (Experimental): Lorcaserin 10 mg tablet each morning and evening
  Interventions: Drug: Lorcaserin 10 mg BID
- Matching Placebo BID (Placebo Comparator): Matching placebo tablet each morning and evening
  Interventions: Drug: Matching Placebo BID

INTERVENTIONS:
Drug: Lorcaserin 10 mg BID — Lorcaserin 10 mg tablet each morning and evening for a duration of 52 or 104 weeks.
  Other Names: APD356
  Arms: Lorcaserin 10 mg BID
Drug: Matching Placebo BID — Matching placebo tablet each morning and evening for a duration of 52 or 104 weeks.
  Arms: Matching Placebo BID

SUMMARY:
The purpose of this study is to assess the weight loss effect of lorcaserin at the end of the first year of treatment (Week 52) and to assess the ability of lorcaserin to maintain weight loss at the end of the second year of treatment (Week 104)

ELIGIBILITY:
Inclusion Criteria:

* Obese adults with a BMI 30 to 45 kg/m2 or overweight adults with a BMI 27 to 29.9 kg/m2 and at least one obesity-related comorbidity (hypertension, dyslipidemia, cardiovascular disease, glucose intolerance, sleep apnea)
* Ability to complete a 2 year study

Exclusion Criteria:

* Diabetes
* Pregnancy
* History of heart valve disease
* Serious or unstable current or past medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3182 (Actual)
Dates: Start 2006-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arena Pharmaceuticals, Inc., San Diego, California, United States

REFERENCES:
- [Derived] Weissman NJ, Smith SR, Fain R, Hall N, Shanahan WR. Effects of lorcaserin on pre-existing valvulopathy: A pooled analysis of phase 3 trials. Obesity (Silver Spring). 2017 Jan;25(1):39-44. doi: 10.1002/oby.21695. Epub 2016 Nov 26. PMID 27888609
- [Derived] Handelsman Y, Fain R, Wang Z, Li X, Fujioka K, Shanahan W. Lorcaserin treatment allows for decreased number needed to treat for weight and glycemic parameters in week 12 responders with >/=5% weight loss. Postgrad Med. 2016 Nov;128(8):740-746. doi: 10.1080/00325481.2016.1240591. Epub 2016 Oct 19. PMID 27659698
- [Derived] Nguyen CT, Zhou S, Shanahan W, Fain R. Lorcaserin in Obese and Overweight Patients Taking Prohibited Serotonergic Agents: A Retrospective Analysis. Clin Ther. 2016 Jun;38(6):1498-1509. doi: 10.1016/j.clinthera.2016.04.004. Epub 2016 May 17. PMID 27206567
- [Derived] Nesto R, Fain R, Li Y, Shanahan W. Evaluation of lorcaserin on progression of prediabetes to type 2 diabetes and reversion to euglycemia. Postgrad Med. 2016 May;128(4):364-70. doi: 10.1080/00325481.2016.1178590. PMID 27116910
- [Derived] Weissman NJ, Sanchez M, Koch GG, Smith SR, Shanahan WR, Anderson CM. Echocardiographic assessment of cardiac valvular regurgitation with lorcaserin from analysis of 3 phase 3 clinical trials. Circ Cardiovasc Imaging. 2013 Jul;6(4):560-7. doi: 10.1161/CIRCIMAGING.112.000128. Epub 2013 May 9. PMID 23661689
- [Derived] Smith SR, Weissman NJ, Anderson CM, Sanchez M, Chuang E, Stubbe S, Bays H, Shanahan WR; Behavioral Modification and Lorcaserin for Overweight and Obesity Management (BLOOM) Study Group. Multicenter, placebo-controlled trial of lorcaserin for weight management. N Engl J Med. 2010 Jul 15;363(3):245-56. doi: 10.1056/NEJMoa0909809. PMID 20647200
- See also: Arena Pharmaceuticals, Inc. Home Page — http://www.arenapharm.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Year 1 - Lorcaserin 10 mg BID: lorcaserin 10 mg BID tablets
- Year 1 - Matching Placebo BID: matching placebo tablets
- Year 2 - Lorc 10 mg BID (Yr 1) / Lorc 10 mg BID (Yr 2): Patients were randomized to lorcaserin in Year 1, completed year 1 study and randomized to lorcaserin in Year 2.
- Year 2 - Lorc 10 mg BID (Yr 1) / Placebo (Yr 2): Patients were randomized to lorcaserin in Year 1, completed year 1 study and randomized to placebo in Year 2.
- Year 2 - Placebo (Yr 1) / Placebo (Yr 2): Patients randomized to placebo in Year 1, completed year 1 and randomized to receive placebo in Year 2.
Period: Year 1
Arm/Group | Year 1 - Lorcaserin 10 mg BID | Year 1 - Matching Placebo BID | Year 2 - Lorc 10 mg BID (Yr 1) / Lorc 10 mg BID (Yr 2) | Year 2 - Lorc 10 mg BID (Yr 1) / Placebo (Yr 2) | Year 2 - Placebo (Yr 1) / Placebo (Yr 2)
Started | 1595 | 1587 | 0 | 0 | 0
Completed | 883 | 716 | 0 | 0 | 0
Not Completed | 712 | 871 | 0 | 0 | 0
Period: Year 2
Arm/Group | Year 1 - Lorcaserin 10 mg BID | Year 1 - Matching Placebo BID | Year 2 - Lorc 10 mg BID (Yr 1) / Lorc 10 mg BID (Yr 2) | Year 2 - Lorc 10 mg BID (Yr 1) / Placebo (Yr 2) | Year 2 - Placebo (Yr 1) / Placebo (Yr 2)
Started | 0 | 0 | 573 | 283 | 697
Completed | 0 | 0 | 426 | 195 | 507
Not Completed | 0 | 0 | 147 | 88 | 190

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Year 1 - Lorcaserin 10 mg BID | Year 1 - Matching Placebo BID | Total
Number analyzed (Participants) | 1593 | 1584 | 3177
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (11.32) | 44.4 (11.11) | 44.1 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1321 | 1331 | 2652
  Male | 272 | 253 | 525

OUTCOME MEASURES:

1. Primary Outcome: Year 1: Co-Primary Endpoint- Proportion (%) of Patients Achieving > or = 5% Weight Loss From Baseline to Week 52
Description: The proportion of patients with a reduction from baseline body weight of 5% or more at the end of year 1.
  Other co-primary endpoints are change from baseline in body weight (kg) at year 1 and the proportion of patients achieving ≥ 10% reduction in body weight at year 1.
Time Frame: 52 weeks
Population: MITT with LOCF
Measure: Number; unit: percentage of participants
Groups:
- Lorcaserin 10 mg BID: lorcaserin 10 mg BID tablets
- Matching Placebo BID: matching placebo tablets
Arm/Group | Lorcaserin 10 mg BID | Matching Placebo BID
Number analyzed (Participants) | 1538 | 1499
percentage of participants | 47.5 | 20.3
Statistical Analysis 1: Comparison: Lorcaserin 10 mg BID vs Matching Placebo BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; Odds Ratio (OR) = 3.6, 95% CI 2-sided [3.0 to 4.2]

2. Primary Outcome: Year 2: Proportion (%) of Patients Maintaining > or = 5% Weight Loss at Week 104
Description: The proportion of patients with a reduction from baseline body weight of 5% or more at the end of year 1 and who maintained this reduction during year 2.
Time Frame: 104 weeks
Population: MITT with LOCF
Measure: Number; unit: percentage of participants
Groups:
- Lorcaserin 10 mg BID (Yr 1) / Lorcaserin 10 mg BID (Yr 2): Patients were randomized to lorcaserin in Year 1, completed year 1 study with a "Responder" status and randomized to lorcaserin in Year 2.
- Lorcaserin 10 mg BID (Yr 1) / Matching Placebo (Yr 2): Patients were randomized to lorcaserin in Year 1, completed year 1 with a "Responder" status and randomized to placebo in Year 2.
Arm/Group | Lorcaserin 10 mg BID (Yr 1) / Lorcaserin 10 mg BID (Yr 2) | Lorcaserin 10 mg BID (Yr 1) / Matching Placebo (Yr 2)
Number analyzed (Participants) | 380 | 175
percentage of participants | 67.9 | 50.3

3. Secondary Outcome: Year 1: Percent Change in Body Weight From Baseline to Week 52
Description: Year 1: The % change in body weight (kg) from baseline to week 52.
Time Frame: 52 weeks
Population: MITT with LOCF
Measure: Least Squares Mean (Standard Error); unit: % change from baseline: body wt (kg)
Arm/Group | Lorcaserin 10 mg BID | Matching Placebo BID
Number analyzed (Participants) | 1538 | 1499
% change from baseline: body wt (kg) | -5.87 (0.18) | -2.20 (0.18)
Statistical Analysis 1: Comparison: Lorcaserin 10 mg BID vs Matching Placebo BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in proportion (%) = -3.67, 95% CI 2-sided [-4.09 to -3.25]

4. Secondary Outcome: Year 2: Percent Change in Body Weight From Week 52 to Week 104
Description: Year 2: The % change in body weight (kg) from week 52 to week 104.
Time Frame: 52 weeks
Population: MITT with LOCF
Measure: Least Squares Mean (Standard Error); unit: % change from baseline: body wt (kg)
Groups:
- Lorcaserin 10 mg BID (Yr 1) / Lorcaserin 10 mg BID (Yr 2): Patients were randomized to lorcaserin in Year 1, completed year 1 study and randomized to lorcaserin in Year 2.
- Lorcaserin 10 mg BID (Yr 1) / Matching Placebo (Yr 2): Patients were randomized to lorcaserin in Year 1, completed year 1 study and randomized to placebo in Year 2.
- Placebo (Yr 1) / Placebo (Yr 2): Patients were randomized to placebo in Year 1 and randomized to placebo in Year 2.
Arm/Group | Lorcaserin 10 mg BID (Yr 1) / Lorcaserin 10 mg BID (Yr 2) | Lorcaserin 10 mg BID (Yr 1) / Matching Placebo (Yr 2) | Placebo (Yr 1) / Placebo (Yr 2)
Number analyzed (Participants) | 553 | 267 | 665
% change from baseline: body wt (kg) | 2.79 (0.23) | 5.38 (0.31) | 1.15 (0.22)
Statistical Analysis 1: Comparison: Lorcaserin 10 mg BID (Yr 1) / Lorcaserin 10 mg BID (Yr 2) vs Lorcaserin 10 mg BID (Yr 1) / Matching Placebo (Yr 2); Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in proportion (%) = -2.58, 95% CI 2-sided [-3.29 to -1.88]
Statistical Analysis 2: Comparison: Lorcaserin 10 mg BID (Yr 1) / Lorcaserin 10 mg BID (Yr 2) vs Placebo (Yr 1) / Placebo (Yr 2); Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in proportion (%) = 1.64, 95% CI 2-sided [1.10 to 2.19]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a period of up to 2 years. The data is separated by group and by year and is inclusive for each year.
Groups:
- Year 2 - Lorc 10 mg BID (Yr 1) / Lorc 10 mg BID (Yr 2): lorcaserin 10 mg BID tablets
- Year 2 - Lorc 10 mg BID (Yr 1) / Matching Placebo (Yr 2): lorcaserin 10 mg BID tablets, matching placebo tablets
- Year 2 - Placebo (Yr 1) / Placebo (Yr 2): matching placebo tablets
Arm/Group | Year 1 - Lorcaserin 10 mg BID | Year 1 - Matching Placebo BID | Year 2 - Lorc 10 mg BID (Yr 1) / Lorc 10 mg BID (Yr 2) | Year 2 - Lorc 10 mg BID (Yr 1) / Matching Placebo (Yr 2) | Year 2 - Placebo (Yr 1) / Placebo (Yr 2)
Serious Adverse Events (participants affected / at risk) | 38/1593 | 37/1584 | 15/573 | 6/283 | 24/697
Other Adverse Events (participants affected / at risk) | 1324/1593 | 1203/1584 | 450/573 | 210/283 | 515/697
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Year 1 - Lorcaserin 10 mg BID (N=1593) | Year 1 - Matching Placebo BID (N=1584) | Year 2 - Lorc 10 mg BID (Yr 1) / Lorc 10 mg BID (Yr 2) (N=573) | Year 2 - Lorc 10 mg BID (Yr 1) / Matching Placebo (Yr 2) (N=283) | Year 2 - Placebo (Yr 1) / Placebo (Yr 2) (N=697)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Breast hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocele (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Giardiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple congenital abnormalities (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (2) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Radiculitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Retinal exudates (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Uterine malposition (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Year 1 - Lorcaserin 10 mg BID (N=1593) | Year 1 - Matching Placebo BID (N=1584) | Year 2 - Lorc 10 mg BID (Yr 1) / Lorc 10 mg BID (Yr 2) (N=573) | Year 2 - Lorc 10 mg BID (Yr 1) / Matching Placebo (Yr 2) (N=283) | Year 2 - Placebo (Yr 1) / Placebo (Yr 2) (N=697)
Arthralgia (Musculoskeletal and connective tissue disorders) | 70 (79) | 75 (87) | 38 (44) | 17 (18) | 43 (51)
Back pain (Musculoskeletal and connective tissue disorders) | 99 (114) | 89 (93) | 34 (39) | 16 (19) | 30 (33)
Constipation (Gastrointestinal disorders) | 106 (116) | 64 (72) | 14 (16) | 8 (9) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 109 (118) | 85 (100) | 34 (38) | 9 (10) | 30 (31)
Dizziness (Nervous system disorders) | 130 (149) | 60 (69) | 10 (11) | 8 (8) | 17 (17)
Dry mouth (Gastrointestinal disorders) | 83 (84) | 37 (37) | 1 (1) | 3 (3) | 2 (2)
Fatigue (General disorders) | 95 (108) | 48 (51) | 15 (15) | 5 (6) | 16 (17)
Gastroenteritis viral (Infections and infestations) | 79 (87) | 64 (67) | 18 (18) | 14 (14) | 21 (25)
Headache (Nervous system disorders) | 287 (388) | 175 (211) | 41 (49) | 18 (25) | 30 (42)
Influenza (Infections and infestations) | 73 (81) | 69 (72) | 38 (39) | 14 (15) | 42 (44)
Nasopharyngitis (Infections and infestations) | 213 (249) | 190 (223) | 94 (114) | 39 (45) | 88 (103)
Nausea (Gastrointestinal disorders) | 119 (141) | 85 (90) | 20 (20) | 9 (9) | 29 (32)
Sinusitis (Infections and infestations) | 114 (139) | 130 (152) | 49 (62) | 30 (33) | 48 (59)
Upper respiratory tract infection (Infections and infestations) | 235 (280) | 189 (216) | 83 (100) | 31 (41) | 112 (131)
Urinary tract infection (Infections and infestations) | 106 (132) | 96 (112) | 41 (48) | 14 (15) | 35 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study results are only allowed with prior written consent from Arena Pharmaceuticals, Inc.